CLINICAL TRIAL: NCT07245225
Title: Acute Effects of High Impact Exercise on Bone Metabolism
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Loughborough University (Other)
Responsible Party: Principal Investigator, Katherine Brooke-Wavell, Professor, Loughborough University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 16204
Record Dates: First submitted 2025-11-14; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Health Adults
Keywords: Exercise; Bone turnover; Extracellular vesicles; Wnt/β-catenin signaling pathway
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm Drop-landing + Control (Experimental): According to the results of random allocation, participants first perform the drop-landing trial, followed by the control trial, with a minimum interval of one week between the two trials.
  Interventions: Behavioral: Exercise
- Arm Control + Drop-landing (Experimental): According to the results of random allocation, participants first perform the control trial, followed by the drop-landing trial, with a minimum interval of one week between the two trials.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — During the drop-landing trial, participants perform drop-landing exercises from a block calibrated to generate approximately four times their body weight in vertical ground reaction force upon landing, employing a stiff-landing technique. Each repetition is separated by a 30-second interval, and 10 repetitions are performed as 1 set, totalling 6 sets. There is a 2-minute rest break between each set, during which the participants are asked to sit on a chair. The entire drop-landing exercise is recorded on the force plate.
  During the control trial, participants are required to walk up and down from the same height block without the requirement to perform the drop-landing movement. The number of repetitions, intervals, and rest breaks are completely consistent with the drop-landing exercise.

SUMMARY:
The goal of this study is to investigate the acute effects of drop-landing exercise on the bone metabolism biomarkers and extracellular vesicles in healthy young males, in order to gain a deeper understanding of the mechanotransduction mechanisms involved in bone metabolism.

The main question aims to answer:

• Does a single bout acute drop-landing exercise change serum sclerostin, other bone signaling markers, and circulating extracellular vesicles levels?

Participants complete both the drop-landing and control trials in a randomized order, with a minimum washout period of one week between trials. During each trial, blood samples are collected at three time points: pre-, immediately post, and 1-hour post drop-landing/control exercise.

ELIGIBILITY:
Inclusion Criteria:

* 18-35 years old
* Healthy
* Male
* Body mass index (BMI) of 18.5-29.9
* Can understand and follow trial instructions

Exclusion Criteria:

* Have any uncontrolled cardiovascular or respiratory disease
* Have severe musculoskeletal or neurological disease likely to affect ability to perform an exercise
* Have medical conditions known to affect musculoskeletal health
* Have medications known to affect bone metabolism (e.g., corticosteroids, thyroxine, antiepileptic, and antiretroviral agents)
* Regular (more than once per week) participation in high-intensity resistance or impact-type exercise in the past 6 months
* Current smoker or vaper

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Serum sclerostin concentration | Blood samples are collected at pre- (baseline), immediately post, 1-hour post drop-landing/control exercise in main trials.
  Serum sclerostin concentration is quantified using an enzyme-linked immunosorbent assay (ELISA) and reported in picograms per milliliter (pg/mL).

SECONDARY OUTCOMES:
Serum dickkopf Wnt signaling pathway inhibitor 1 (DKK1) concentration | Blood samples are collected at pre- (baseline), immediately post, 1-hour post drop-landing/control exercise in main trials.
  Serum DKK1 concentration is quantified using an enzyme-linked immunosorbent assay (ELISA) and reported in picograms per milliliter (pg/mL).
Serum osteoprotegerin (OPG) concentration | Blood samples are collected at pre- (baseline), immediately post, 1-hour post drop-landing/control exercise in main trials.
  Serum OPG concentration is quantified using an enzyme-linked immunosorbent assay (ELISA) and reported in picograms per milliliter (pg/mL).
Serum irisin concentration | Blood samples are collected at pre- (baseline), immediately post, 1-hour post drop-landing/control exercise in main trials.
  Serum irisin concentration is quantified using an enzyme-linked immunosorbent assay (ELISA) and reported in picograms per milliliter (pg/mL).
Circulating extracellular vesicle (EV) particle concentration and size | Blood samples are collected at pre- (baseline), immediately post, 1-hour post drop-landing/control exercise in main trials.
  EVs are isolated from plasma using ultracentrifugation. EV particle concentration is quantified by nanoparticle tracking analysis (NTA) and reported as particles per milliliter (particles/mL). EV size is also assessed by NTA and reported in nanometers (nm).
Ground reaction force during drop-landing exercise | Ground reaction force is recorded during each drop-landing exercise.
  Ground reaction force is recorded in newtons (N) during each drop-landing exercise using a force plate in the drop-landing trial. Ground reaction force is reported in multiples of body weight (×BW).

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Brooke-Wavell, Principal Investigator — Loughborough University
Locations (1):
- Loughborough University, Loughborough, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Once the analysis is complete and the planned analyses are published, the investigators will consider sharing anonymized IPD upon request, subject to the necessary agreements.